CLINICAL TRIAL: NCT04940754
Title: Ankle Arthrodesis Nail Combined With Locking Compression Plate to Stabilize Two-level Pathologic Tibial Fractures
Brief Title: Ankle Arthrodesis Nail for 2-level Pathologic Tibial Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Orthopaedie Zentrum Zuerich (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUE
Record Dates: First submitted 2021-06-10; First posted 2021-06-28 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Bone Metastases; Fracture Nonunion; Bone Lesion
Keywords: fragility fracture, old age
MeSH Terms: conditions — Fractures, Ununited | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: Use of an approved implant for expanded application
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stabilzation of Fracture (Other): Arthrodesis nail used for stabilzation of a fracture, single patient
  Interventions: Procedure: osteosynthesis

INTERVENTIONS:
Procedure: osteosynthesis — Closed reduction, internal fixation

SUMMARY:
Tibial pseudarthrosis in 83 year old patient suffering from pathologic fractures

DETAILED DESCRIPTION:
The arthrodesis nail for hind foot problems is used as salvage for tibial fractures after failed plate fixation,

ELIGIBILITY:
Inclusion Criteria:

- old age, fragility fracture, tibia

Exclusion Criteria:

* active osteomyelitis

Ages: 80 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-04-08 (Estimated); Study Completion 2022-05-08 (Estimated)

PRIMARY OUTCOMES:
Weight bearing tolerance | 1 year
  Measuring walking distance

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedie Zentrum Zuerich, Zurich, Switzerland